CLINICAL TRIAL: NCT00247806
Title: Prevalence of Lactose Intolerance Following Stem Cell Transplantation in Pediatric Patients.
Brief Title: Prevalence of Lactose Intolerance Following Stem Cell Transplantation
Status: Terminated | Type: Observational
Why Stopped: Too few patients completed the study once enrolled.
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Colin C Barker, University of British Columbia
Other Study IDs: C05-0180
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2005-10

CONDITIONS: Lactose Intolerance
Keywords: Pilot, pediatric, stem cell transplant, lactose intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
It is currently assumed that all patients are lactose intolerant post bone marrow transplantation. This pilot study is to assess what the incidence of lactose intolerance is after bone marrow transplantation in children. This will be done using a lactose breath test.

DETAILED DESCRIPTION:
All pediatric patients over the age of 4 years who are scheduled for a stem cell transplant will be approached to assess whether what the incidence of lactose intolerance is in the post transplant period and how quickly recovery occurs. A baseline lactose and lactulose breath test will be performed followed by repeat lactose breath tests starting 2 weeks after day 0 and repeated every fortnight for 10 weeks. Stool pH and reducing substances will be checked at the time of the breath tests to see if there is any correlation.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned to undergo a stem cell transplant.

Exclusion Criteria:

* Refusal to participate
* Unable to perform breath tests on request (generally under the age of 4 years.)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Barker, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada